CLINICAL TRIAL: NCT02946411
Title: Correlation of Hospital Stay Length With the Glucose Measured Continuously Levels After Cardiac Surgery
Brief Title: Correlation of Hospital Stay Length With the Glucose Levels After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2016-785.080
Record Dates: First submitted 2016-10-20; First posted 2016-10-27 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Stress Hyperglycemia
Keywords: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: The glucose of 48 patients will be measured during 5 days after cardiac surgery.
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Glucose level will be measured after cardiac surgery.

SUMMARY:
The study is designed to test if there is any correlation between the glucose levels in the postoperatory period and the length of hospital stay.

DETAILED DESCRIPTION:
The stress hyperglycemia commonly observed in the postoperatory period, there have been several studies to assess if there is benefit of having a strict glucose control or not.

This study will assess if there is correlation between the glucose levels measured continuously with the length of the stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Physical status classification of the American Society of Anesthesiologists (ASA) II-IV
* Patients programmed for cardiac surgery
* Any body mass index

Exclusion Criteria:

* Pregnant women
* Chronic Kidney Disease (CKD) Stage 2 or higher

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a programmed cardiac surgery
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Glucose | 5 days
  Glucose will be continuously monitored for 5 days

SECONDARY OUTCOMES:
Hospital stay | [Days] Within the first 20 days after surgery
  The days that the patient remains in the hospital after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gallardo, Dr., Principal Investigator — Investigator
Locations (1):
- Hospital de cardiología, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided